CLINICAL TRIAL: NCT00758290
Title: Clinical Study to Evaluate Dental Plaque
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP- Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2008-PLA-13-RR
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Triclosan; Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Triclosan/Fluoride
- B (Experimental)
  Interventions: Drug: Fluoride/triclosan

INTERVENTIONS:
Drug: Triclosan/Fluoride — Brush twice daily for 3 weeks
  Arms: A
Drug: Fluoride/triclosan — Brush daily for 3 weeks
  Arms: B

SUMMARY:
Clinical research study to determine anti-plaque efficacy of a prototype toothpastes for a 3 week brushing regiment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers at least 20 - 51 years of age
* Good general health
* Must sign informed consent form
* Minimum of 15 natural uncrowned teeth (excluding third molars) must be present
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form
* Medical condition which requires pre-medication prior to dental visits/procedures
* Moderate or advanced periodontal disease or heavy dental tartar (calculus)
* 5 or more decayed untreated dental sites at screening (cavities)
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that are currently affecting salivary function
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1
* Pregnant or nursing women
* Participation in any other clinical study within 1 week prior to enrollment into this study
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates
* Current use of Antibiotics for any purpose
* Presence of an orthodontic appliance which interferes with plaque scoring
* History of allergy to common toothpaste ingredients
* History of allergy to arginine (amino acid)
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 20 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Corby, DDS, Principal Investigator
Locations (1):
- Bluestone Center for Clinical Research, NYU College of Dentistry, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Period: Overall Study
Arm/Group | Fluoride/Triclosan | Triclosan/Fluoride
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride/Triclosan | Triclosan/Fluoride | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants] — Twenty four panelists were enrolled, but 1 was discontinued due to non-compliance with study visits. Twenty three panelists comleted study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 12 | 23
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.5 (11.7) | 30.3 (7.1) | 31.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Index
Description: Plaque units measured on a scale between 0 to 5. No plaque=0;5=2/3 of tooth covered in plaque
Time Frame: 4 Day
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride/Triclosan | Triclosan/Fluoride
Number analyzed (Participants) | 12 | 12
Units on a scale | 2.48 (0.34) | 2.42 (0.39)
Statistical Analysis 1: Comparison: Fluoride/Triclosan vs Triclosan/Fluoride; Test type: Superiority or Other; p = 0.05, ANOVA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days